CLINICAL TRIAL: NCT00001987
Title: Natural History of Disorders of Insulin Resistance
Brief Title: Genetic Studies of Insulin and Diabetes
Status: Recruiting | Type: Observational
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 760006; 76-DK-0006
Record Dates: First submitted 2000-01-28; First posted 2000-01-31 (Estimated); Last update posted 2026-01-13 (Actual); Status verified 2026-01-09

CONDITIONS: Diabetes Mellitus; Severe Insulin Resistance
Keywords: Diabetes Mellitus; Severe Insulin Resistance; Type B Insulin Resistance; Natural History
MeSH Terms: conditions — Diabetes Mellitus; Insulin Resistance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (2):
- Healthy Volunteers: Healthy Volunteers
  Interventions: Device: HR-pQCT scan
- Patients with severe insulin resistance: patients with severe insulin resistance manifesting with acanthosis nigricans, hyperinsulinemia, type A and B insulin resistance syndromes, and patients with lipodystrophy.
  Interventions: Device: HR-pQCT scan

INTERVENTIONS:
Device: HR-pQCT scan — HR-pQCT is a non-invasive, low-dose three-dimensional imaging method used to evaluate volumetric bone mineral density and bone microarchitecture of peripheral skeletal sites, including distal radius and distal tibia. HR-pQCT has an ability to differentiate between cortical and trabecular bone compartments providing density and structure parameters.

SUMMARY:
The study will allow researchers to obtain blood, plasma, DNA, and RNA for genetic studies of insulin. There will be a focus on the causes of insulin resistance and diabetes mellitus. Insulin is a hormone found in the body that controls the level of sugar in the blood. Insulin resistance refers to conditions like diabetes when insulin does not work properly. In this study researchers would like to compare patients with diabetes and other forms of insulin resistance to normal individuals. The study will investigate how insulin attaches to cells.

Researchers will take 4 to 6 ounces (100-150 ml) of blood from adult patients and may request up to 12 ounces (one unit) of blood if necessary. Skin samples may be taken for a biopsy if further genetic testing is necessary. In addition some patients may be asked not to eat for up to 72 hours prior to testing.

DETAILED DESCRIPTION:
Study Description:

Insulin is the key hormone responsible for regulating the level of glucose in plasma. In several disease states (e.g., obesity, type 2 diabetes, and acromegaly), the target cells are resistant to insulin action. Insulin resistance leads to metabolic complications including diabetes, dyslipidemia, cardiovascular disease, non-alcoholic fatty liver disease, and reproductive dysfunction. The intramural research program of the NIDDK has a long history of studying patients with rare disorders of extreme insulin resistance. We use what is learned from these rare patients both to develop therapeutics for rare diseases, and to apply what is learned to understand more common forms of insulin resistance.

Objectives:

Primary Objectives: (1) To understand the pathophysiology of insulin resistance and its relationship to diabetes, dyslipidemia, cardiovascular disease, liver disease, kidney disease, reproductive function, bone disease, and other organ dysfunction, (2) To study the molecular genetics underlying various causes of insulin resistance and diabetes mellitus, (3) To understand the natural history of insulin resistance disorders, including their response to FDA approved therapies, and (4) To conduct ex vivo studies of the physiology and pathophysiology underlying disorders of insulin resistance, and possible treatments for these disorders, using cells and tissues collected in this study.

Endpoints:

Primary Endpoint: Genetic causes of insulin resistance

Secondary Endpoints: Diabetes control (hemoglobin A1c) and complications (rates of micro- and macrovascular disease)

ELIGIBILITY:
* INCLUSION CRITERIA:

Three categories of subjects will be included in this study:

* Patients with evidence for insulin resistance or a disorder associated with severe insulin resistance, including:

  * Patients with various syndromes of lipodystrophy
  * Patients with known or suspected mutations on the insulin receptor gene
  * Patients with known or suspected autoantibodies to the insulin receptor
  * Patients with other severe forms of insulin resistance
* Family members of patients, above
* Healthy control subjects without insulin resistance

Inclusion criteria for each group of subjects are given below:

* Patients with evidence for severe insulin resistance or a disorder associated with severe insulin resistance must meet all of the following criteria:

  * Suspected severe insulin resistance, or a disorder associated with severe insulin resistance, as evidenced by one or more of the following:
  * Hyperinsulinemia (i.e. fasting insulin >30microU/mL)
  * High insulin requirement (> 2 units per kg per day or > 200 units total per day)
  * Phenotypic features suggesting a defect in glucose/lipid metabolism:

    * Acanthosis nigricans
    * Lipodystrophy/abnormal fat distribution
    * Xanthomata
    * Fatty liver
  * Known or suspected mutations of the insulin receptor gene
  * Known or suspected autoantibodies to the insulin receptor
  * Age >= 6 months
  * Ability of subject or Legally Authorized Representative (LAR) to understand and the willingness to sign a written informed consent document.
* Family members of patients, above (either affected or unaffected) must meet all of the following criteria:

  * Biological relatives of patients in category (1) in whom a genetic cause of insulin resistance is known or suspected.
  * Age >= 6 months
  * Ability of subject (and/or legal guardian, for minor subjects) to understand and the willingness to sign a written informed assent/consent document.
* Healthy control subjects Cohort 1 must meet all of the following criteria.

  * Ability of subject (and/or legal guardian, for minor subjects) to understand and the willingness to sign a written informed assent/consent document.
  * In good general health with no known active medical conditions as evidenced by medical history
  * Age >= 12 years
* Healthy control subjects Cohort 2. Subjects from Cohort 1 may be included in Cohort 2 if they meet the following ADDITIONAL inclusion criteria.

  * Fasting glucose <100 mg/dL
  * HbA1c <5.7%
  * Fasting triglycerides <150 mg/dL
  * Fasting insulin <30 mcU/mL
  * BMI <27 kg/m^2 or <90th percentile for age/sex (whichever is lower)

EXCLUSION CRITERIA:

* Patients with evidence for insulin resistance or a disorder associated with severe insulin resistance

  --none
* Family members of patients, above

  --Pregnant at the time of enrollment
* Healthy control subjects Cohort 1

  * Current use of prescription or non-prescription medication. Certain exceptions are permitted, including topical medications, vitamins, and hormonal contraceptives. Other medications may be permitted at the discretion of the investigators.
  * Recent (past 2 months) use of drugs or supplements that alter glucose or lipid metabolism (e.g. niacin, fish oil, red yeast rice)
  * History of diabetes or abnormal glucose tolerance
  * Psychiatric or cognitive disorder that will, in the opinion of the investigators, limit the subject's ability to provide informed consent/assent, or to comply with study procedures
  * Pregnant or lactating
* Healthy control subjects Cohort 2. Subjects from Cohort 1 may NOT be included in Cohort 2 if they have any of the following ADDITIONAL exclusion criteria.

  * Abnormal screening labs, including the following:

    * ALT or AST more than 1.5 times the upper limit of normal
    * Glycosuria
    * Clinically significant anemia
    * Low eGFR (<60 mL/min/1.73m^2)
    * Any other abnormality that, in the opinion of the investigator, will increase risk to the subject from participation, or interfere with interpretation of study data

Ages: 6 Months to 120 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Subjects with severe insulin resistance disorders.
Sampling Method: Non-Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 1976-02-01 (Actual)

PRIMARY OUTCOMES:
Diabetes control | every 6-12 months
  To help prevent additional health issues associated with poor glucose and insulin levels.
Genetics of insulin resistance | End of Study
  To discover the cause of the insulin resistance to better assist with treatment for it.
Pathophysiology of insulin resistance and its relationship to cardiovascular disease. | End of study
  To understand the pathophysiology of insulin resistance and its relationship to cardiovascular disease.
Obtain tissue samples for ex vivo studies. | End of study
  To understand physiology and pathophysiology of insulin resistance and develop possible treatments.

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca J Brown, M.D., Principal Investigator — National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No
Subject level data will be shared upon request after appropriate collaboration agreements are in place.

REFERENCES:
- [Derived] Okawa MC, Tuska RM, Lightbourne M, Abel BS, Walter M, Dai Y, Cochran E, Brown RJ. Insulin Signaling Through the Insulin Receptor Increases Linear Growth Through Effects on Bone and the GH-IGF-1 Axis. J Clin Endocrinol Metab. 2023 Dec 21;109(1):e96-e106. doi: 10.1210/clinem/dgad491. PMID 37595266
- [Derived] Walzer D, Turcu AF, Jha S, Abel BS, Auchus RJ, Merke DP, Brown RJ. Excess 11-Oxygenated Androgens in Women With Severe Insulin Resistance Are Mediated by Adrenal Insulin Receptor Signaling. J Clin Endocrinol Metab. 2022 Aug 18;107(9):2626-2635. doi: 10.1210/clinem/dgac365. PMID 35696182
- [Derived] Okawa MC, Cochran E, Lightbourne M, Brown RJ. Long-Term Effects of Metreleptin in Rabson-Mendenhall Syndrome on Glycemia, Growth, and Kidney Function. J Clin Endocrinol Metab. 2022 Feb 17;107(3):e1032-e1046. doi: 10.1210/clinem/dgab782. PMID 34718628
- [Derived] Meral R, Malandrino N, Walter M, Neidert AH, Muniyappa R, Oral EA, Brown RJ. Endogenous Leptin Concentrations Poorly Predict Metreleptin Response in Patients With Partial Lipodystrophy. J Clin Endocrinol Metab. 2022 Mar 24;107(4):e1739-e1751. doi: 10.1210/clinem/dgab760. PMID 34677608
- [Derived] Nguyen ML, Sachdev V, Burklow TR, Li W, Startzell M, Auh S, Brown RJ. Leptin Attenuates Cardiac Hypertrophy in Patients With Generalized Lipodystrophy. J Clin Endocrinol Metab. 2021 Oct 21;106(11):e4327-e4339. doi: 10.1210/clinem/dgab499. PMID 34223895
- [Derived] Sekizkardes H, Chung ST, Chacko S, Haymond MW, Startzell M, Walter M, Walter PJ, Lightbourne M, Brown RJ. Free fatty acid processing diverges in human pathologic insulin resistance conditions. J Clin Invest. 2020 Jul 1;130(7):3592-3602. doi: 10.1172/JCI135431. PMID 32191645
- [Derived] Klubo-Gwiezdzinska J, Lange M, Cochran E, Semple RK, Gewert C, Brown RJ, Gorden P. Combined Immunosuppressive Therapy Induces Remission in Patients With Severe Type B Insulin Resistance: A Prospective Cohort Study. Diabetes Care. 2018 Nov;41(11):2353-2360. doi: 10.2337/dc18-0884. Epub 2018 Sep 10. PMID 30201849
- [Derived] Brown RJ, Joseph J, Cochran E, Gewert C, Semple R, Gorden P. Type B Insulin Resistance Masquerading as Ovarian Hyperthecosis. J Clin Endocrinol Metab. 2017 Jun 1;102(6):1789-1791. doi: 10.1210/jc.2016-3674. PMID 27911591
- [Derived] Kassai A, Muniyappa R, Levenson AE, Walter MF, Abel BS, Ring M, Taylor SI, Biddinger SB, Skarulis MC, Gorden P, Brown RJ. Effect of Leptin Administration on Circulating Apolipoprotein CIII levels in Patients With Lipodystrophy. J Clin Endocrinol Metab. 2016 Apr;101(4):1790-7. doi: 10.1210/jc.2015-3891. Epub 2016 Feb 22. PMID 26900642
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_1976-DK-0006.html